CLINICAL TRIAL: NCT01789216
Title: Improving Pain Management and Long Term Outcomes Following High Energy Orthopedic Trauma (Pain Study)
Acronym: PAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: W81XWH1020090
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Orthopaedic Fractures
Keywords: Pilon fractures; Calcaneus fractures; Acute pain; Chronic pain; Isolated; unilateral; Grade I; Grade II; open; closed
MeSH Terms: conditions — Acute Pain; Chronic Pain; Lymphoma, Follicular | interventions — Anti-Inflammatory Agents, Non-Steroidal; Meloxicam; Ketorolac; Ketorolac Tromethamine; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Standard pain management + perioperative intravenous placebo & oral placebo.
  Control group will receive an oral dose of placebo up to two hours prior to surgery and twice daily for up to 48 hours following any surgery, in addition to an intravenous dose of placebo up to two hours prior to surgery and every 6 hours for up to 48 hours following surgery. All study medications will be in addition to standard of care pain medication.
  *Previous preoperative protocol was removed due to difficulty of medication adherence and limited importance of preoperative regimen to the intervention overall.
  Interventions: Drug: placebo
- NSAID (Active Comparator): Standard pain management + perioperative intravenous ketorolac & oral placebo.
  The NSAID group will receive 30 mg of intravenous (IV) ketorolac (Ketorolac 30 mg/ml dose vial, NDC 00409-3795-01; manufacturer: Hospira) administered up to two hours prior to the procedure and every 6 hours for up to 48 hours following the procedure. In addition, as part of the perioperative protocol, patients will receive an oral dose of placebo up to two hours prior to the procedure and every 12 hours for up to 48 hours following the procedure.
  *Previous preoperative protocol was removed due to difficulty of medication adherence and limited importance of preoperative regimen to the intervention overall.
  Interventions: Drug: NSAID
- Gabapentinoid (Active Comparator): Standard pain management + perioperative intravenous placebo & oral pregabalin.
  The Pregabalin group will receive an oral bolus dose of 300 mg of pregabalin up to two hours prior to the procedure and a 75 mg dose every 12 hours for up to 48 hours following the procedure. In addition, as part of the perioperative protocol, patients will receive an IV dose of placebo up to two hours prior to the procedure and every 6 hours for up to 48 hours following the procedure.
  *Previous preoperative protocol was removed due to difficulty of medication adherence and limited importance of preoperative regimen to the intervention overall.
  Interventions: Drug: Gabapentinoids

INTERVENTIONS:
Drug: NSAID
  Other Names: Meloxicam/Mobic (NDC 68382-000-01; manufacturer: Zydus; encapsulated in size AA; empty capsule shells, backfilled with Avicel by Fisher Clinical Services (Bristol); LLC); Ketorolac/Toradol (NDC 00409-3795-01; manufacturer: Hospira)
  Arms: NSAID
Drug: Gabapentinoids
  Other Names: Pregablin/Lyrica (NDC 00071-1014-68; manufacturer: Pfizer; encapsulated in size; AA empty capsule shells, backfilled with Avicel by Fisher Clinical Services; (Bristol) LLC,; Lyrica, NDC 00071-1018-68; manufacturer: Pfizer; encapsulated; in size AA empty capsule shells, backfilled with Avicel by Fisher Clinical; Services (Bristol) LLC)
  Arms: Gabapentinoid
Drug: placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to definitively resolve questions regarding the use of multimodal pharmacologic pain management for orthopedic trauma patients in the context of a multicenter, randomized clinical trial.

Also, as a significant proportion of this population develops chronic post traumatic osteoarthritis (PTOA), a sub-objective of this study is to examine the etiology and incidence of chronic pain and PTOA in this population.

DETAILED DESCRIPTION:
In this study, will test whether adjunctive analgesic therapy during the pre and peri-operative period, in addition to standard of care pain management, can improve overall pain control and pain related outcomes without increasing analgesic related side effects.

Patients will be randomized into three treatment groups. The intervention will begin within 48 hours of admission and continue for up to the time of definitive fixation.

Group 1: standard pain management, plus intravenous and oral placebo for up to 48 hours following definitive fixation.

Group 2: standard pain management, plus intravenous NSAIDs (ketorolac) and oral placebo for up to 48 hours following definitive fixation.

Group 3: standard pain management, plus intravenous placebo and oral pregabalin for up to 48 hours following definitive fixation.

Specific Aim 1: Evaluate the effect of standard pain management (Group 1) vs. standard pain management plus peri-operative NSAIDs (Group 2 - meloxicam + ketorolac) in the treatment of severe limb fractures.

Hypothesis 1a: When compared to patients who received standard of care pain management, patients treated with NSAIDs will: (1) have reduced post operative opioid utilization; (2) report reduced levels of persistent pain; and (3) have noninferior rates of surgery for nonunion.

Hypothesis 1b: When compared to patients who received standard of care pain management, patients treated with NSAIDs will benefit from (1) improved post operative pain control; (2) improved pre operative pain control; (3) reduced lengths of stay; (4) reduced pain interference; (5) improved functional outcomes; (6) lower levels of depression and post-traumatic stress disorder (PTSD); (7) improved overall health status; and (8) have noninferior rates of analgesic treatment related side effects.

Specific Aim 2: Evaluate the effect of standard pain management (Group 1) vs. standard pain management plus pre and peri-operative pregabalin (Group 3) in the treatment of severe limb fractures.

Hypothesis2a : When compared to patients who received standard of care pain management, patients treated with pregabalin will: (1) have reduced post operative opioid utilization; (2) report reduced levels of persistent pain; and (3) have noninferior rates of surgery for nonunion.

Hypothesis 2b: When compared to patients who received standard of care pain management, patients treated with pregabalin will benefit from (1) improved post operative pain control; (2) improved pre operative pain control; (3) reduced lengths of stay; (4) reduced pain interference; (5) improved functional outcomes; (6) lower levels of depression and post-traumatic stress disorder (PTSD); (7) improved overall health status; and (8) have noninferior rates of analgesic treatment related side effects.

Specific Aim 3: Estimate the incremental cost effectiveness of each adjunctive analgesic therapy relative to standard of care analgesic therapy in the treatment of severe limb fractures. Costs will be estimated from both the health care provider perspective and the societal perspective. The time horizon for cost-effectiveness analysis will be based on the actual period of observation. Incremental cost-effectiveness ratios will be calculated for: (a) study group 2 (NSAIDS - meloxicam + ketorolac) relative to standard of care; and (b) study group 3 (pregabalin) relative to standard of care. For purpose of cost-effectiveness analysis, the effect will be measured as unit change in specific outcome metrics at up to 15 months (or longer period as available) compared to baseline. The following cost-effectiveness metrics, all relative to standard of care, will be reported:

1. incremental cost per unit change in the Brief Pain Inventory
2. incremental cost per unit change in the Short Muscular Function Assessment (SFMA)
3. incremental cost per unit change in health state preference ("utility") as derived from the VR-12.

PTOA Pilot Study: Additional funding was received from NIH to conduct a pilot, observational study of post-traumatic osteoarthritis (PTOA), leveraging current resources of the Pain study. PTOA is an important outcome in the population to be enrolled in the Pain study. The aims of the PTOA Study are to: (1) measure the incidence of PTOA and chronic pain for up to 24 months following fracture reduction surgery and (2) quantify the extent to which fracture severity and post-reduction contact stress are related to the development of PTOA. Accomplishment of these aims will require (1) for all patients with ankle fractures in the Pain study: complete a PTOA survey at 12 months and at any subsequent visits that are conducted as part of standard of care and provide access to all standard of care imaging studies completed during the study period and (2) for a subset of 60 pilon fracture patients enrolled in the Pain study for whom post-operative CT scans are not standard of care, obtain additional consent for completion of a study-funded post-operative CT scan and 24 month radiographic study

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following types of injuries:

   1. Unilateral, Grade I &II open or closed pilon (distal tibial plafond), calcaneus, talus fractures and Lisfranc dislocations requiring operative treatment with fixation; or
   2. Unilateral, open (type I, II, or IIIA) ankle fractures with associated dislocation on presentation (OTA 44B3 or 44C) requiring operative treatment with fixation; or
   3. Unilateral, open or closed distal and proximal humerus (OTA 11A-C and OTA 13 A-C); or
   4. Open femoral shaft fracture (OTA 32 A-C; Gustilo Type I-IIIC) or open or closed supracondylar femur fractures (OTA 33 A-C); or
   5. Open or closed tibial plateau or shaft fractures (OTA 42 A-C or 43 A-C)
   6. Any combination of the above injuries which are surgically treated as a whole
2. Patients who present to the admitting hospital acutely or clinic following an initial assessment in the Emergency Department, for care up to 10 days following initial injury.
3. Patients 18-80 years old inclusive.
4. Patients who are English or Spanish competent.
5. Treating physicians agree that none of the study drugs are indicated for standard of care treatment for this patient.
6. Patients able to be followed at the METRC facility for at least 12 months following injury.

Exclusion Criteria:

1. Patients unable to provide informed consent.
2. Patients with chronic pain being presently treated with opioid or gabapentinoid prescription or any other alternative therapy.
3. Patients who are current IVDA
4. Patients with bilateral or ipsilateral injuries requiring surgery
5. Patients with other orthopedic or non-orthopedic injuries requiring operative intervention
6. Patients with severe osteopenia.
7. Patients who are skeletally immature (defined as less than 18 years of age or no radiographic evidence of epiphyseal closure).
8. Patients who are expected to have a post-surgical stay less than 24 hours.
9. Patients with a history of allergy to any drugs in the study.
10. Patients unable to swallow oral medications or without adequately functioning GI tract.
11. Patients with a history of gastrointestinal bleeds or gastric perforation.
12. Patients with a history of stroke or heart attack.
13. Patients currently receiving an aspirin or NSAID regimen (exception: low dose (81 mg) aspirin. See section 6.5) Patients with any bleeding disorders.
14. Patients with severe renal failure. Patients with moderate renal failure may participate in the study at a modified dose. See Section 9.6.
15. Patients undergoing daily treatment with systemic glucocorticoids before surgery.
16. Patients using angiotensin-converting enzyme (ACE) inhibitors, who may be at increased risk of developing angioedema with pregabalin.
17. Patients likely to have severe problems maintaining follow-up, including patients diagnosed with a severe psychiatric conditions, patients who live too far outside the hospital's catchment area, patients who are incarcerated and patients who have unstable housing situations.
18. Patients who experienced a loss of consciousness consistent with a clinical diagnosis of a closed head injury, or concern of a cerebrovascular bleed secondary to traumatic brain injury.
19. Patients with a GCS <15
20. Patient speaks neither English nor Spanish.
21. Patients who are pregnant or lactating at time of screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Opioid Utilization | 1 year
  Morphine equivalent opioid utilization during initial hospitalization through 48 hours following definitive fixation.
Persistent Pain | 1 year
  Patient reported persistent pain states at standard of care visits 3, 6 and 12 months following hospital discharge. Measured using the Brief Pain Inventory (BPI) and an additional battery of questions to assess neuropathic pain (painDETECT).
Surgery for non-union | 1 year
  Defined as non-prophylactic surgery for nonunion performed between six months and a year following initial hospital discharge.

SECONDARY OUTCOMES:
Post Surgical Pain Intensity | 2 days
  Pain intensity at 12-hour intervals during the 48 hours following definitive fixation surgery. Abstracted from medical record and supplemented by participant pain logs. At least one time point will be assessed using the Multidimensional Post Surgical Pain Scale in order to study multiple pain dimensions.
Pre Surgical Pain Intensity | 2 days
  Pain intensity at 12-hour intervals between study enrollment and definitive fixation surgery. Abstracted from medical record and supplemented by participant pain logs.
Length of Index Hospitalization | 1 year
  Defined as the hospitalization during which the definitive fixation occurs. Length of stay for all other study injury related hospitalizations will also be abstracted.
Adverse Effects and Complications | 2-3 weeks
  Will include nonunion, wound closure complications, bleeding complications (particularly perioperative bleeding due to loss of platelet function and gastrointestinal bleeding), as well as pain treatment related adverse effects. These include nausea, vomiting, constipation, sedation, pruritis, respiratory depression, somnolence, dizziness, headaches, coordination problems, peripheral edema, blurred vision, gastrointestinal symptoms and irritation, renal impairment, platelet inhibition, angioedema, and post operative delirium. Adverse effects and complications will be assessed by both patient report of symptoms during the period between enrollment and 48 hours post definitive fixation, and by clinical survey of symptoms during index hospitalization and at discharge from additional surgical admissions up to definitive fixation.
Functional Outcome | 1 year
  The SMFA (Short Musculoskeletal Function Assessment) is a shorter version of the 101-item Musculoskeletal Function Assessment (MFA) questionnaire. The SMFA is a 46-item questionnaire consisting of the dysfunction index and the bother index. The dysfunction index has 34 items for assessment of patient function, while the bother index consists of 12 items designed to detect how much patients are bothered by functional items. The SMFA has been evaluated for reliability, validity and responsiveness in trauma populations. To be assessed at 6 and 12 months.
Generic Health Status | 1 year
  The generic health status will be measured by the VR-12 instrument from which a VR-6D can be computed for the purpose of a cost-utility analysis. The VR-12 is a multipurpose self-administered generic measure of health status. It was developed to measure health-related quality of life, estimate disease burden and compare disease-specific benchmarks across populations. The VR-12 items measure eight health domains: general health perceptions; physical functioning; role limitations due to physical and emotional problems; bodily pain; energy-fatigue, social functioning and mental health. The instrument produces a physical health and mental health summary measure. To be assessed at 6 and 12 months.
Depressive Symptoms | 1 year
  The presence of depressive symptoms will be measured using the nine item depression scale of the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a well validated tool for assisting clinicians in diagnosing depression. There are two components of the PHQ-9: (1) assessing symptoms and functional impairment to make a tentative depression diagnosis, and (2) deriving a severity score. The PHQ-9 is based directly on the diagnostic criteria for major depressive disorder in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV). To be assessed at 12 months.
Post Traumatic Stress (PTSD) | 1 year
  PTSD will be measured using the standard PTSD Checklist (PCL), a 17-item measure that elicits responses for each of the DSM-IV disorders that comprise the diagnostic criteria for PTSD (intrusive, avoidant, and arousal symptoms). The psychometric properties of the PCL have been well established and it is the most widely used measure of PTSD. Both civilian and military versions are available. The military version will be used for all those patients on active duty at the time of their injury. To be assessed at 12 months.
Medical Costs | 1 year
  Costs for the index hospitalization and subsequent hospitalizations (within one year) will be derived using hospital bills, outpatient bills and professional fees. Hospital costs will be calculated from charges at the revenue center/cost department line level using cost-to-charge ratios (CCRs) computed from the hospital-specific Medicare Cost Reports. Billing data will be supplemented or imputed by identifying medical resource utilization as documented in study case report forms, categorizing resources using standard medical billing codes, and assigning costs based on Medicare fee schedules. Of particular interest will be resource utilization and costs associated with the index hospital admission, surgical procedures for bone grafting and nonunion, subsequent admissions for complications, and post-operative follow-up care.
Fracture Severity | 1-2 years
  Fracture severity will be measured using standard of care CT scans. In severe fractures, this image will be obtained after application of a temporary joint spanning external fixator. Thus, the fracture severity analysis will be based on fractured distal tibias with limb alignment provisionally controlled. After definitive fracture reconstruction, a second CT scan will be obtained at the 3 month follow up time point, for assessment of chronic contact stress challenge. The second CT scan will be obtained for all patients for whom it is standard of care.
Fracture Classification | 1-2 years
  Fracture classification will be obtained using radiographs of the patient's injured ankle at presentation and after each surgical intervention according to standard of care practice. These radiographs will be used for clinical care, to classify the fractures, and at follow-up to assess outcome. Radiographs will be obtained at the time of initial hospital evaluation, immediately following treatment and at follow up clinic visits according to standard of care. Final clinical assessments and radiographs will be obtained as close to 12 months as routine practice allows. At practices where patients are routinely followed for more than 12 months and 24 month clinical assessments and radiographs will be conducted, at which point all study-related activities will be completed. A subset of 60 patients, identified prospectively, will provide an additional CT 3 months following definitive fixation, and will provide a final set of radiographs 24 months following definitive fixation.

OTHER OUTCOMES:
PTOA sub-study assessment | 1-2 years
  Among patients in the Pain study, data relevant to the development of PTOA will be collected observationally. All radiographic images, including CT scans and x-rays, taken per standard of care in the first year will be obtained. Additionally, for those patients routinely receiving follow-up beyond 12 months, weight bearing radiographs of the ankle taken at between one and two years after injury will be used to assess and characterize the development of PTOA. In the subset of 60 pilon fracture patients actively recruited into the PTOA pilot study, CT scans following definitive fixation, all radiographic images taken per standard of care, in addition to a final set of weight bearing radiographs of the ankle taken at 24 months will be used to assess and characterize the development of PTOA. The presence of PTOA will be determined using the Kellgren and Lawrence (KL) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Renan Castillo, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Lawrence Marsh, MD, Principal Investigator — University of Iowa Hospitals & Clinics; Katherine Frey, RN, MPH, MS, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (17):
- United States (17):
  - University of Miami Ryder Trauma Center, Miami, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Eskenazi Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland, R Adams Cowley Shock Trauma Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Carolinas Medical Center, Charlotte, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - UT Health: The University of Texas Health Science Center at Houston Medical School, Houston, Texas
  - Naval Medical Center Portsmouth, Portsmouth, Virginia